CLINICAL TRIAL: NCT05560867
Title: Neural Mechanisms of Motor Recovery With Technology Assisted Training for Post-stroke Hemiparesis
Brief Title: Neural Mechanisms of Motor Recovery With Technology Assisted Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues with study robotics preventing completion of the research intervention
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robynne Braun, MD, PhD, Assistant Professor, Department of Neurology, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00093740
Record Dates: First submitted 2022-07-25; First posted 2022-09-29 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hemiparesis; Stroke Sequelae
Keywords: stroke; robot-assisted rehabilitation; neural networks; fnirs; rehabilitation
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patient Robot-Assisted Training Group (Other): Patients will undergo robot-assisted physical therapy three times a week, for a total of 9 sessions, while functional near-infrared spectroscopy data is collected.
  Interventions: Device: robot-assisted training

INTERVENTIONS:
Device: robot-assisted training — These training platforms use gamified training tasks to improve motor control in the hemiparetic arm
  Other Names: IMT InMotion Wrist Robot; IMT InMotion2 Shoulder-Elbow Robot; IMT InMotion2 Planar Robot

SUMMARY:
Stroke is a leading cause of disability that often impairs arm function and activities of daily living. The costs of rehabilitation are significant and practical constraints often limit therapy to the first few months after stroke. However many studies have shown that patients in the later stages post-stroke can still continue to benefit from rehabilitation. Technology-assisted therapy may offer a means to efficiently provide ongoing therapies to patients in the later stages (>6 months) post-stroke. This study will determine which patients are best able to benefit from this therapy approach, and will also expand our knowledge of which brain structures need to be intact for patients to benefit from technology-assisted training. The results of this study will help to improve rehabilitation and quality of life for disabled Americans.

DETAILED DESCRIPTION:
Study Description: This study will investigate the neural mechanisms of technology-assisted-training for post-stroke hemiparesis by using functional near-infrared-spectroscopy (fNIRS). Patients with hemiparesis affecting the arm will be brought in for 3 weeks of technology-assisted-training while having fNIRS recordings of their brain activity. Analysis of these brain activation patterns will help determine what areas of the brain are necessary to respond to this type of training.

Objectives: 1) to investigate brain network activity changes that occur during technology-assisted-training and 2) to determine the baseline residual brain network connectivity required for patients to respond to robot-assisted-training.

Endpoints: The study will evaluate increases in cortical connectivity between bilateral primary motor areas, angular gyrus and parietal operculum to test the hypothesis that cortical connectivity in these areas will positively correlate with improvement in technology-assisted-assessments. The study will also assess baseline connectivity of the angular gyrus and parietal operculum to sensorimotor networks to test the hypothesis that cortical connectivity in these areas will predict reductions in arm motor impairments that occur with technology-assisted-training.

Study Population: Patients of either gender with chronic (at least 6 months or more) hemiparesis of the arm caused by a single unilateral stroke will be recruited from Baltimore city and the surrounding counties.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 88 years
* Able to provide informed consent based on Evaluation to Sign Informed Consent.
* History of clinically defined, unilateral hemiparetic stroke, with radiologic exclusion of other possible diagnosis, causing weakness in 1 arm 6 months or more prior to enrollment.
* Fugl-Meyer upper extremity score <= 50 at time of enrollment
* Medically stable to participate in the study and have mobility, visual, and cognitive abilities sufficient to follow directions and engage in the gamified therapeutic tasks.

Exclusion Criteria:

* Undergoing any significant medical treatments requiring regular visits, treatments, or therapies at the time of enrollment or anytime during the study.
* Hair or scalp implant that would not allow near infrared spectroscopy probes to sit on scalp.
* Injection of botulinum toxin to the paretic arm within 3 months of enrollment or during the study or injection of daxibotulinumtoxinA within 6 months of enrollment or during the study
* Orthopedic, rheumatologic, or other medical disease that would make the procedures of participation dangerous, painful, or uncomfortable.
* Contraindications to MRI, including intracranial magnetic items, implanted pumps, pacemakers, or stimulators, or claustrophobia.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in cortical connectivity measures as assessed using MRI | Baseline MRI will be collected at the time of study enrollment (for a total of up to 4 weeks during study enrollment)
  Cortical connectivity is assessed between bilateral primary motor areas, angular gyrus and parietal operculum. MRI sequences include T1 MPRAGE, BOLD (T2*), FLAIR T2, ASL, and DTI.
Changes in cortical connectivity measures as assessed using fNIRS | Baseline fNIRS collected at the time of study enrollment, with repeated fNIRS measures at each therapy treatment session (for a total of up to 4 weeks during study enrollment)
  Cortical connectivity is assessed between bilateral primary motor areas, angular gyrus and parietal operculum.

SECONDARY OUTCOMES:
Changes in arm kinematics (position) | Baseline kinematics at the time of study enrollment with repeated measures at each therapy treatment session (for a total of up to 4 weeks during study enrollment)
  Arm kinematics measures of position collected by the rehabilitation training technology devices
Changes in arm kinematics (velocity) | Baseline kinematics at the time of study enrollment with repeated measures at each therapy treatment session (for a total of up to 4 weeks during study enrollment)
  Arm kinematics measures of velocity collected by the rehabilitation training technology devices
Changes in arm kinematics (acceleration) | Baseline kinematics at the time of study enrollment with repeated measures at each therapy treatment session (for a total of up to 4 weeks during study enrollment)
  Arm kinematics measures of acceleration collected by the rehabilitation training technology devices
Changes in Fugl-Myer Scores for the Upper Extremity ("FM-UE") | At the time of enrollment with repeated measures at each therapy treatment session (for a total of up to 4 weeks during study enrollment)
  Standardized bedside test examining the degree of motor impairment for the arm/hand. Scores range from 0 - 66 with higher scores representing better recovery.
Changes in Action Research Arm Test | At the time of enrollment (pre-training) with a second measure at the final study session (post-training) (for a total of up to 4 weeks during study enrollment).
  Standardized bedside test examining behavioral tasks for the arm/hand. Scores range from 0-57 points, with a maximum score of 57 points indicating better performance.
Changes in Wolf Motor Function Test ("WMFT") | At the time of enrollment (pre-training) with a second measure at the final study session (post-training) (for a total of up to 4 weeks during study enrollment).
  Standardized bedside test examining behavioral tasks for the arm/hand. Score Ranges Minimum 0 to Maximum 75; Lower scores are indicative of lower functioning levels.
Changes in Shoulder Abduction Finger Extension ("SAFE") score | At the time of enrollment with repeated measures at each therapy treatment session (for a total of up to 4 weeks during study enrollment)
  Standardized bedside test examining strength of the arm/hand. Scores range from 0-10 with higher scores representing better strength.
Changes in NIH Stroke Scale Score ("NIHSS") | At the time of enrollment with repeated measures at each therapy treatment session (for a total of up to 4 weeks during study enrollment)
  Standardized bedside test to assess stroke symptoms. Scores range from 0 - 42, where higher scores indicate greater symptom severity.
Changes in Stroke Impact Scale ("SIS") | At the time of enrollment (pre-training) with a second measure at the final study session (post-training) (for a total of up to 4 weeks during study enrollment)
  Standardized questionnaire examining patient perceptions of how stroke impacts their function and quality of life. Scores range from 0 to 100 with higher scores indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No